CLINICAL TRIAL: NCT01243125
Title: A Multicenter, Double-blind, Crossover Design, Pilot Study to Evaluate the Effect of NVC-422 Catheter Irrigation on Urinary Catheter Patency
Brief Title: Study to Evaluate NVC-422 for Urinary Catheter Blockage and Encrustation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovaBay Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CL1001
Record Dates: First submitted 2010-11-15; First posted 2010-11-18 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Urinary Catheter Blockage and Encrustation
Keywords: Blockage; Encrustation; Catheter; Spinal Cord Injury; SCI
MeSH Terms: conditions — Spinal Cord Injuries | interventions — NVC-422; Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVC-422 (Experimental)
  Interventions: Drug: NVC-422, 0.2%
- Saline (Placebo Comparator)
  Interventions: Drug: Sterile normal saline, 0.9%

INTERVENTIONS:
Drug: NVC-422, 0.2% — 0.2% NVC-422 (sterile), 25 ml instilled and retained in catheter for 15 min, 2x/day; 8 treatments administered over a 26 day period
  Other Names: N,N-dichloro-2,2-dimethyltaurine
  Arms: NVC-422
Drug: Sterile normal saline, 0.9% — Saline (sterile), 25 ml instilled and retained in catheter for 15 min, 2x/day; 8 treatments administered over a 26 day period
  Other Names: 0.9% Sodium chloride for injection, USP
  Arms: Saline

SUMMARY:
NVC-422 is a topical, non-antibiotic, fast-acting, broad-spectrum anti-microbial, which exhibits the potential to prevent the growth of urinary pathogens, including Proteus and others.

The use of a catheter irrigation solution that can prevent biofilm formation and encrustation leading to blockage may keep the catheter patent longer, resulting in fewer catheter changes, potentially lower incidence of UTIs, and better patient quality of life.

The study population will include male and female spinal cord injury (SCI) and other neurogenic bladder patients with chronic indwelling transurethral urinary catheters who have a recent repeated history of urinary catheter encrustation and/or blockage.

Subjects will receive two treatment regimens: one treatment regimen with NVC-422 sterile irrigation solution and one treatment regimen with sterile saline irrigation solution. Each treatment regimen will consist of a total of 8 treatments, with a washout period between treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury (SCI) or other neurogenic bladder patient requiring a chronic indwelling urinary catheter with history of catheter blockage and/or encrustation
* Screening within 30 days of first treatment

Exclusion Criteria:

* Systemic antibiotics within 7 days of first treatment
* Investigational drug or device within 30 days of enrollment
* Current infection that requires treatment with systemic antibiotics
* Recent history of significant autonomic dysreflexia (requiring intervention or treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Catheter patency following treatment | 26 days
  Cross sectional area (percent of open area that is not encrusted) will be determined at pre-selected loci on the catheter

SECONDARY OUTCOMES:
Incidence of catheter blockage requiring early removal | 26 days
  Catheters removed prior to completion of treatment regimen will be assessed for each treatment group
Assessment of biofilm of catheter | 26 days
  Qualitative and quantitative assessment of biofilm of catheter will be determined for all catheters removed
Assessment of encrustation of catheter | 26 days
  Qualitative and quantitative assessment of encrustation of catheter will be determined for all catheters removed

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D. Krantz, MD, PhD, Study Director — NovaBay Pharmaceuticals / kkrantz@novabaypharma.com
Locations (8):
- United States (8):
  - Los Amigos Research and Education Institute (LAREI), Downey, California
  - Specialists in Urology, Naples, Florida
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - Integrity Medical Research, Mountlake Terrace, Washington